CLINICAL TRIAL: NCT06863909
Title: Study on the Effectiveness of Journaling as an add-on to Cognitive Behavioral Therapy: A Randomized Controlled Trial
Brief Title: Study on the Effectiveness of Journaling as an add-on to Cognitive Behavioral Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 611/2024BO2
Record Dates: First submitted 2025-02-19; First posted 2025-03-07 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-02

CONDITIONS: Affective Disorders; Rumination; Childhood Trauma; Eating Disorder; Substance Use Disorder; Personality Disorder; Mental Disorder
MeSH Terms: conditions — Mood Disorders; Rumination Syndrome; Feeding and Eating Disorders; Substance-Related Disorders; Personality Disorders; Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A total of 80 patients will be included, and they will be assigned to one of two treatment groups: one group will receive standard treatment, while the second group will receive additional tasks/techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Treatment as Usual (TAU)
- Treatment as usual + Journaling (Experimental)
  Interventions: Behavioral: Journaling; Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Journaling — In the journaling condition, participants will be asked to keep a therapy journal twice a day in addition to the content of the cognitve behavioral therapy. At the beginning of the day, patients are to set a daily goal that aligns with their therapy goals (e.g., remaining calm when negative thoughts arise), and at the end of the day, they will reflect on the day itself and the work done on their therapy goals.
  Arms: Treatment as usual + Journaling
Behavioral: Treatment as Usual (TAU) — Patients in this arm receive standard treatment (cognitive behavioral therapy) for their individual diagnosis. The study participation spans a period of 24 sessions (short-term psychotherapy KZT1&2), during which the severity of symptoms will be assessed at the beginning of each session (duration approx. 2 minutes). Additionally, participants will be asked to answer some questions about basic documentation (diagnoses, symptoms) at the beginning and end of the study (duration approx. 20 minutes).

SUMMARY:
The aim of the present study is to examine the effects of keeping a therapy journal (journaling) on the effectiveness of cognitive behavioral therapy (CBT). Homework assignments are a fundamental component of behavioral therapies. In line with the learning theory foundation of behavioral therapies, various types of homework are used to facilitate learning processes between therapy sessions and to enable patients to make progress. One way to enhance individual goal setting and reflection in patients is through the use of "therapy journals."

The goal of the planned project is to evaluate the effectiveness of goal-oriented journal writing as an additional element in cognitive behavioral therapy (CBT). To do this, N = 80 psychotherapy patients will be randomly assigned to two treatment groups: CBT vs. CBT + Journaling.

DETAILED DESCRIPTION:
As part of this study, the investigators are examining the effectiveness of certain therapeutic techniques that could improve the effectiveness of psychotherapy. A total of 80 patients will be studied, and they will be assigned to one of two treatment groups: one group will receive standard treatment, while the second group will receive additional tasks/techniques. The study will span a period of 24 sessions (short-term psychotherapy KZT1&2), during which the severity of their symptoms will be assessed at the beginning of each session (duration approx. 2 minutes). Additionally, participants will be asked to answer some questions about basic documentation (diagnoses, symptoms) at the beginning and end of the study (duration approx. 20 minutes).

The investigators assure that the personal data they collect will be protected in accordance with the European Data Protection Regulation. Collected data will only be analyzed in anonymized form, meaning without mentioning any names, and may be published in scientific journals. All data will be stored in encrypted form using personal codes. All data will be digitally archived for a period of 10 years on a well-secured drive at the University Hospital Tübingen; only the study leaders (Dr. Rosenbaum and Dr. Ehlis) are authorized to re-identify the data. The investigators would like to inform that the collected data will not be used for diagnostic purposes regarding possible pathological changes. There are no health risks associated with this study, and while it is unlikely to benefit personally from it, the participation will contribute to scientific knowledge.

ELIGIBILITY:
Inclusion Criteria:

* patients in ambulant cognitive behavioral therapy

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire for the Evaluation of Psychotherapy Progress (german: Fragebogen zur Evaluation von Psychotherapieverläufen (english translation: Questionnaire for evaluating the course of psychotherapy) (FEP-2)) | From enrollment to the end of treatment at 24 weeks
  Number of patients exhibiting reliable changes in FEP-2 scores between baseline and end of treatment.
  FEP-2 = Fragebogen zur Evaluation von Psychotherapieverläufen (english translation: Questionnaire for evaluating the course of psychotherapy). Minimum = 1; Maximum = 5. Higher scores mean a better outcome.
Questionnaire for the Evaluation of Psychotherapy Progress (german: Fragebogen zur Evaluation von Psychotherapieverläufen (english translation: Questionnaire for evaluating the course of psychotherapy)(FEP-2)) | From enrollment to the end of treatment at 24 weeks
  Number of sessions until patients exhibit reliable changes in FEP-2 scores between baseline and end of treatment.
  FEP-2 = Fragebogen zur Evaluation von Psychotherapieverläufen (english translation: Questionnaire for evaluating the course of psychotherapy). Minimum = 1; Maximum = 5. Higher scores mean a better outcome.
Questionnaire for the Evaluation of Psychotherapy Progress (german: Fragebogen zur Evaluation von Psychotherapieverläufen (english translation: Questionnaire for evaluating the course of psychotherapy)(FEP-2)) | From enrollment to the end of treatment at 24 weeks
  Investigation of the changes in FEP-2 scores between the groups between baseline and end of treatment.
  FEP-2 = Fragebogen zur Evaluation von Psychotherapieverläufen (english translation: Questionnaire for evaluating the course of psychotherapy). Minimum = 1; Maximum = 5. Higher scores mean a better outcome.
Questionnaire for the Evaluation of Psychotherapy Progress (german: Fragebogen zur Evaluation von Psychotherapieverläufen (english translation: Questionnaire for evaluating the course of psychotherapy)(FEP-2)) | From enrollment to the end of treatment at 24 weeks
  Investigation of a repeated-measures ANOVA to compare the mean FEP2 values (intent-to-treat; last observation carried forward) across different phases: baseline (sessions 1-5), early change (sessions 6-15), and late change (sessions 15-25).
  FEP-2 = Fragebogen zur Evaluation von Psychotherapieverläufen (english translation: Questionnaire for evaluating the course of psychotherapy). Minimum = 1; Maximum = 5. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Number of days patients completed the diary | From enrollment to the end of treatment at 24 weeks
  At the end of each therapy session, the therapist assesses the frequency with which the diary was completed as an indicator of the complicance of the patient.
  The "frequency of completion" is measured in the number of days in which the diary was completed (e.g. diary was completed on 5 days = 5). The maximum of the scale is calculated by the number of days that have passed since the last session. Higher scores mean a better outcome.
Custom questionnaire: Quality of implementation of goals | From enrollment to the end of treatment at 24 weeks
  At the end of each therapy session, the therapist rates the quality of the implementation of the goals as an indicator of the compliance of the patient.
  The scale "Quality of implementation of goals" is measured on a custom 5-point Likert scale. The therapist rates:
  1. = did not implement the rules of goal setting on any day
  2. = implemented the rules of goal setting on less than half of the days, but not never
  3. = implemented the rules of goal setting on half of the days
  4. = implemented the rules of goal setting on more than half of the days, but not always
  5. = implemented the rules of goal setting every day The minimum is correspondingly 1, the maximum 5. Higher scores mean a better outcome.
Custom questionnaire: Quality of reflection | From enrollment to the end of treatment at 24 weeks
  At the end of each therapy session, the therapist rates the quality of the reflection as an indicator of the compliance of the patient.
  The scale "Quality of reflection" is measured on a custom 5-point Likert scale. The therapist rates:
  1. = not reflected on any day if necessary
  2. = reflected on less than half of the days, but not never, if necessary
  3. = reflected on half of the days if necessary
  4. = reflected on more than half of the days, but not always, if necessary
  5. = reflected on every day if necessary The minimum is correspondingly 1, the maximum 5. Higher scores mean a better outcome.
Custom questionnaire: Quality and quantity of homework completion | From enrollment to the end of treatment at 24 weeks
  At the end of each therapy session, the therapist rates the quality of the overall quality and quantity of the homework completion.
  This scale is measured on a custom 5-point Likert scale. The therapist rates:
  1. = not at all
  2. = a little
  3. = moderate
  4. = good
  5. = very good The minimum is correspondingly 1, the maximum 5. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Christine Ehlis, Dr., Principal Investigator — University Hospital Tübingen Department of Psychiatry and Psychotherapy
Locations (1):
- University Hospital Tübingen, Department of Psychiatry and Psychotherapy, Tübingen, Germany